CLINICAL TRIAL: NCT03844958
Title: Effect of Consuming Red Furu On Serum Vitamin B12, Homocysteine And Other Cardio-Metabolic Risk Factors In Healthy Young Volunteers: A Randomized Controlled Trial
Brief Title: Effect of Red Furu Consumption on Serum Vitamin B12 and Homocysteine Concentration In Healthy Young Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhejiang University T.T
Record Dates: First submitted 2019-02-02; First posted 2019-02-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Red furu; Metabolism; Randomized
MeSH Terms: interventions — Soy Foods

STUDY DESIGN:
Intervention Model Description: The study will apply the parallel method and volunteers will be randomized into two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Furu (Experimental): Volunteer was randomized into group red furu
  Interventions: Other: Red Furu; Other: Tofu
- Fresh Tofu (Experimental): Volunteer was randomized into group tofu
  Interventions: Other: Red Furu; Other: Tofu

INTERVENTIONS:
Other: Red Furu — 50 g red furu was consumed with 2 slices of plain bread for one-day
  50 g Fresh tofu was consumed with 2 slices of plain bread for one-day
Other: Tofu — 50 g Fresh tofu was consumed with 2 slices of plain bread for one-day
  50 g red furu was consumed with 2 slices of plain bread for one-day

SUMMARY:
The aim of the present study is to investigate the effect of red furu (Chinese fermented soybean product) consumption on serum vitamin B12, Homocysteine concentration and other cardio-metabolic risk factors in healthy young volunteers.

DETAILED DESCRIPTION:
The study will apply the parallel study method and participants will be randomized into two groups. In the randomized controlled clinical trial, twenty-three healthy young volunteers (11 females and 12 males, aged 19-39 years) were recruited from Zhejiang University, China. They were randomly assigned to two groups of either red furu (n=11, 5 females and 6 males) or tofu (n=12, 6 females and 6 males). Volunteers consumed a provided meal, either 50 g of red furu or tofu with two slices of bread for 1 day breakfast meal. Volunteers also recorded their normal dietary intake during the 3 days trial period using provided self-report food diary. Fasting blood sample was drawn at 0h, 24h and 72h. Serum VB12, Hcy and other cardio-metabolic risk factors were measured by standard methods.

Test Meals:

Red Furu Group: 50 g of red furu with 2 slices of bread. Tofu Group: 50 g of plain tofu eaten with 2 slices of bread. Volunteers will refrain from consumption of fermented products 1 week prior to the study. Thereafter subject feed on control diet and intervention diet for 1 day. Volunteers' normal diets and test meals will be recorded on a self-administered questionnaire, followed by testing serum vitamin B12, Homocysteine and other biochemical parameters.

5-10 mL blood will be collected per session. Blood will be collected: 3 times (0h-24h-72h).Participants will be asked to fast for 10-12 hours prior to the blood draw.

ELIGIBILITY:
Inclusion Criteria:

* 20-39 Years
* All Races

Exclusion Criteria:

* Taking antibiotics or vitamin B12 supplements within 1 month prior to enrollment

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Serum Vitamin B12 | 0-24-72 Hours
  Serum vitamin B12 concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Serum Homocysteine | 0-24-72 Hours
  Serum homocysteine concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd

SECONDARY OUTCOMES:
Serum Folate | 0-24-72 Hours
  Serum folate concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Serum Iron | 0-24-72 Hours
  Serum iron concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Serum Ferritin | 0-24-72 Hours
  Serum ferritin concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Glucose | 0-24-72 Hours
  Serum glucose concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Total cholesterol | 0-24-72 Hours
  Serum total cholesterol concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Triglyceride | 0-24-72 Hours
  Triglyceride concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
High-density cholesterol | 0-24-72 Hours
  High-density cholesterol concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd
Low-density cholesterol | 0-24-72 Hours
  Low-density cholesterol concentration was measured by a clinical chemistry analyzer by Hangzhou Golden Field Medical Laboratory Co., Ltd

OTHER OUTCOMES:
Normal Dietary Nutrient Intake | 0-24-72 Hours
  Calculated at Zhejiang University by the researcher using the Chinese Food Software

CONTACTS AND LOCATIONS:
Overall Officials: Duo Li, Doctor, Study Director — Zhejiang University
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Han BZ, Rombouts FM, Nout MJ. A Chinese fermented soybean food. Int J Food Microbiol. 2001 Apr 11;65(1-2):1-10. doi: 10.1016/s0168-1605(00)00523-7. PMID 11322691
- [Background] Kwak CS, Lee MS, Oh SI, Park SC. Discovery of novel sources of vitamin b(12) in traditional korean foods from nutritional surveys of centenarians. Curr Gerontol Geriatr Res. 2010;2010:374897. doi: 10.1155/2010/374897. Epub 2011 Mar 8. PMID 21436999
- [Background] Xu L, Du B, Xu B. A systematic, comparative study on the beneficial health components and antioxidant activities of commercially fermented soy products marketed in China. Food Chem. 2015 May 1;174:202-13. doi: 10.1016/j.foodchem.2014.11.014. Epub 2014 Nov 8. PMID 25529671